CLINICAL TRIAL: NCT06371963
Title: The Relative Energy Deficiency in Sports (REDs) in Swedish Athletes Study
Brief Title: Relative Energy Deficiency in Sports (REDs) in Swedish Athletes
Acronym: REDs-Sweden
Status: Completed | Type: Observational
Sponsor: Linnaeus University (Other)
Collaborators: Swedish Olympic Committee (Unknown); Swedish Research Council for Sport Science (Other); World Anti-Doping Agency (Other)
Responsible Party: Principal Investigator, Anna Melin, Professor, Linnaeus University
Other Study IDs: LinnaeusU REDs
Record Dates: First submitted 2024-02-26; First posted 2024-04-17 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-05

CONDITIONS: RED S; Eating Disorders
Keywords: Observational study; REDs; Eating disorders; Cross-sectional study; Elite athletes; Sweden; Physiological assessments; Performance; Microbiota; Immune function; Resting metabolic rate; Energy availability; Biomarkers; Reproductive dysfunction; The biological passport; Exercise addiction; Gastrointestinal function
MeSH Terms: conditions — Relative Energy Deficiency in Sport; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Gut microbiota composition bacterial DNA from fecal samples,whole blood, serum (only eligible elite athletes participating in physiological testing, anticipated n=44).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Elite Athletes: Senior Swedish male and female national team and recruiting squad athletes.
- Gender and age matched controls: Healthy male and female non-elite athletic controls.

SUMMARY:
Background: Relative Energy Deficiency in Sport (REDs) describes impairment of health and performance due to problematic (long-term/severe) low energy availability (LEA), with or without eating disorders. LEA is frequently reported in sports with high training volumes, especially in leanness demanding sports, and 20% of female and 9% of male Norwegian national team athletes have been reported to have eating disorders. Potential trigger factors are e.g., dieting, injuries, coaching behavior, and subculture aspects e.g., focus on low body weight. The main questions that will be addressed are: 1. What is the prevalence of eating disorders and REDs among Swedish elite athletes and controls? 2. What is the impact of problematic LEA on health and performance aspects in both male and female athletes? Methods: National team athletes and gender and matched controls will be invited to an anonymous on-line survey. Elite athletes who agree to participate, will be invited to assessment of eating disorders, nutritional and physiological status (e.g., metabolic and endocrine markers, bone health, microbiota, dietary intake, energy availability, and performance).

DETAILED DESCRIPTION:
The syndrome of REDs describes impairment of physiological functions e.g., reproduction and bone health with negative impact on performance. The etiology behind is problematic low energy availability (LEA), defined as low energy intake relative to exercise energy expenditure relative to fat free mass. Eating disorders can either proceed or result from REDs. LEA induces metabolic and endocrine alterations, and energy balance at a lower level prevents further weight-loss. Therefore, most athletes with LEA have a body weight within the normal range, and low resting metabolic rate is a recognized LEA surrogate marker.

LEA suppresses anabolic hormones e.g. estradiol/testosterone, while cortisol levels increase, and bone formation markers are reduced. Low testosterone levels have been reported in male endurance athletes, with potential negative effects on fertility. Among Irish male athletes from different sports 23% were identified with low libido and associated with increased injury risk. Menstrual disturbances due to LEA is frequently reported, and is associated with low bone mineral density and injuries.

Glucose is an important substrate for the muscles and an essential substrate for brain neurons and immune cells. Low glucose availability is considered a major trigger to the alterations of the hypothalamic-pituitary axis hormones causing suppression of the sex and thyroid hormones and increase in cortisol. Blood glucose homeostasis is therefore protected with several mechanism (hepatic gluconeogenesis, increased lipolysis and ketogenesis) during prolonged LEA. Hence, hypoglycemia is a marker of a prolonged and severe catabolic state.

LEA has been associated with gastrointestinal problems in female athletes, derived from hormonal and dietary factors affecting motility and digestion. Long-term LEA in patients with anorexia nervosa is associated with profound alterations of the gut microbiome, with negative impact on gastrointestinal function and immunologic processes, and a reduced microbial diversity is therefore suggested as a potential useful biomarker of REDs in athletes. It is therefore relevant to investigate the associations between the gut microbiome, Gastrointestinal function and immunology status in athletes with and without clinical indication of LEA.

LEA affects both men and women, athletes as well as recreational active people however, the threshold and endocrine response seem to differ between gender. Although menstrual disturbances has been frequently reported in female athletes for decades, few studies have investigated the impact on performance, and no study has yet investigated the performance effects of low libido in male athletes. Furthermore, no study has investigated microbial diversity in male and female athletes with clinical symptoms of LEA. Therefore, it is highly relevant to investigate aspects of physiology, nutrition, performance, and sport environment regarding REDs and eating disorders in both male and females.

Objective: The aims of the study are to investigate the prevalence of athletes at risk of eating disorders and REDs among Swedish athletes and controls, and to investigate physiological aspects of elite athletes with and without problematic LEA. Furthermore, to investigate if there is a difference in nutritional status (metabolic and endocrine markers, iron- vitamin D status, energy availability, glucose homeostasis, resting metabolic rate, body composition including bone mineral density), gut microbiota (including associations to immunity), immune function, and performance, in athletes diagnosed with REDs according the International Olympic Committee REDs Clinical Assessment Tool vs. gender matched athletes without REDs. An additional aim is to evaluate if problematic LEA affects biological markers in the biological passport also called "Athlete Biological Passport" in anti-doping.

Methodology and plan of work National senior team and recruiting squad athletes from Swedish sport federations will be invited to an anonymous on-line survey. The 20 minute on-line survey includes: Eating Disorder Examination Questionnaire (EDE-Q). An EDE-Q global score ≥ 2.3 for females and ≥ 1.68 for males indicate risk of EDs; Exercise Addiction Inventory (EAI). A total EAI-score 24-30 indicate compulsive exercise; LEA in Females Questionnaire (LEAF-Q) and LEA in Males Questionnaire (LEAM-Q) to categorize athletes ar risk of LEA; Major Depression Inventory (MDI) to detect depression symptoms; Swedish Acceptance and Action Questionnaire (SAAQ) to assess psychological flexibility; and Motivation to Change Questionnaire (MCQ) to asses the ability for behavioral changes.

Participants who are interested in participating in an on-line diagnostic eating disorder examination interview (the EDE-16) and/or physiological testing, provide their name, cell-phone number, and e-mail address after completing the online survey, and will thereafter be invited to the sport physiology lab for the next phase of the study (physiological assessments).

On the day of the physiological examination, the participants will be asked to deliver a fecal sample. Gut microbiota composition bacterial DNA will be sequenced using next-generation sequencing of microbial genes.

Fasting resting metabolic rate will be measured, using a ventilated open hood system. The ration between measured and predicted resting metabolic will be calculated, and low resting metabolic rate will be defined as resting metabolic rate ratio < 0.90.

Blood samples will be collected and stored (-80°) for later analyses according to standard laboratory procedures (e.g. iron- and vitamin D status, hormones, metabolic, bone and immune markers).

Body weight, height (fixed stadiometer), fat free mass, fat mass and bone mineral density (whole body, femur, and lumbar spine) will be measured using dual-energy x-ray absorptiometry. Low bone mineral density will be defined as Z score -1 to -2 in at least one measured site and osteoporosis as Z-score ≤-2.

After a standardized meal and warm up, a bicycle ergometer exercise test will be performed (6 minutes at 50 watt, followed by 12-14 watt per minute increased workload until exhaustion). Heart rate and an air-tight mask covering the mouth and nose will be used to measure peak oxygen uptake. Capillary lactate will be drawn before, direct after and 5 minutes after the test. Explosive lower body power will be assessed through a counter movement jump-test. Isometric mid-thigh pull will be performed to assess whole body strength and force production. A Wingate-test will be performed to assess muscular power and anaerobic capacity. Post exercise blood-samples will be drawn and stored (-80°) for later analyses according to standard laboratory procedures (e.g., immune markers).

Participants will be asked to wear a subcutaneous continuous blood glucose monitor, an accelerometer, throughout the day except during training where they will wear heart rate monitors and register all training sessions in their home environment for 7 consecutive days. During 4 days in the the same period they will be asked to register all food intake using an electronic kitchen scale and an on-line nutrient program while information of energy and nutrient intake is blinded for the participants. Energy and nutrient intake will be calculated using a nutrient analysis program. Training heart rate and training logs will be used to assess exercise energy expenditure based on individual prediction equations from measured heart rate and corresponding energy expenditure during the peak oxygen uptake test. Energy availability will be calculated by subtracting mean exercise energy expenditure from mean energy intake relative to fat free mass.

Eumenorrheic athletes will be tested on day 2-6 of menstruation, while other athletes will be tested when convenient. All materials (electronic kitchen scale, heart rate monitor, fecal sample collective tube and a prepaid security envelops for returning materials) will be provided.

The skills and equipment for all assessments are available at the Linnaeus University including preparation, storage, and analysis of blood. Fecal samples will be analyzed at the Department of Nutrition, Exercise and Sport, University of Copenhagen.

Power calculation: to provide 80% power to detect a clinically relevant difference in sex hormones a minimum of 14 females (estradiol standard deviation 79.0 nmol/L) and 8 males (total testosterone standard deviation 7.4 pmol/L) in each group will be included.

Recruitment will be performed via the Swedish Olympic Committee, the national sport federations, and social media. The on-line surveys will be launched via the REDs Sweden project webpage and will be open March 2023 to June 2024. Recruitment of age and gender matched controls to the online survey will be performed via social media. Athletes who agree to participate in physiological testing will be continuously scheduled for tests and assessments.

Ethical reviews: The study will follow the checklist issued by the national committees for research ethics and the Helsinki Declaration. Ethical approval has been approved (2021-07031-01). All information and results will be coded (anonymized) before analysis and stored according the general data protection regulation. A list with codes connecting participant names and information will be kept safely locked in by the principal investigator at the Linnaeus University. There are no expected risks with participation. The radiation during the Dual-energy X-ray absorptiometry measurement is negligible. Participants may feel uncomfortable during the assessment of resting metabolic rate and blood sampling. The study collaborators will make sure that participants feel safe during all measurements. If a diagnosis is identified, participants will be referred to the health care system. Participants will be informed regarding ethical rights, the project, expected time cost for participation, and feedback on individual results.

ELIGIBILITY:
Inclusion:

* National-team level athletes
* Non-elite athletic controls

Exclusion (physical assessment):

* chronic illness (e.g., diabetes, hypothyroidism)
* injury
* smoking
* pregnancy
* hormonal contraceptive use

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Swedish male and female national team athletes and gender- and age matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Self-reported eating disorders | Day one
  Participants: Female and male elite athletes and age and gender matched controls.
  An on-line version of the Eating Disorder Examination Questionnaire (EDE-Q) will be used comprising of 28 items, 4 sub-scales (restrained eating, eating-, body-, and weight concerns), and a global score. An EDE-Q global score ≥ 2.3 for females and ≥1.7 for males indicate risk of eating disorder.

SECONDARY OUTCOMES:
Eating disorders | Through study completion, an average of 1 year
  Participants: Elite athlete and controls.
  Diagnostic interview using the eating disorder examination (EDE-16).
Self-reported reproductive function in females not using hormonal contraceptives | Day one
  Participants: Elite athletes and controls.
  The Low Energy Availability in Females Questionnaire (LEAF-Q) comprises 25 items divided into 4 variables: 1) gastrointestinal symptoms, 2) injuries, 3) hormonal contracptives and 4) menstrual function that are scored on a Likert scale (0-46). The higher the score the higher risk of gastrointestinal dysfunction, injuries and menstrual dysfunction.
  Menstrual cycle lengths ≥ 21 days and ≤ 35 days resulting in 9 or more consecutive periods per year indicate eumenorrhea plus results from outcome 4.
  Primary amenorrhea: No menarche by age 15 years Oligomenorrhea: menstrual cycle length > 35 days plus results from outcome 4. Secondary amenorrhea: absence of ≥ 3 consecutive menstrual bleedings. No menarche or no menstrual bleeding the last 3 months plus results from outcome 4.
Reproductive function in females not using hormonal contraceptives | Through study completion, an average of 1 year
  Participants: Female elite athletes (n=28).
  Eumenorrhea: evidence of luteinizing hormone surge, and estrogen, androgen and prolactin levels within normal reference range plus correct categorization by outcome 3.
  Oligomenorrhea and secondary amenorrhea: androgens and prolactin levels within normal reference range plus correct categorization from outcome 3.
Self-reported reproductive function in males | Day one
  Participants: Elite athletes and controls.
  Low Energy Availability in Males Questionnaire (LEAM-Q) comprising of 4 items regarding libido. A low sex drive score is generated by using scores equal or greater than 2 on "Sex drive in general" or equal or greater than 2 on "The number of morning erections" and equal or greater than 1 for "Morning erections compared to normal" to represent reproductive dysfunction plus results from outcome 6.
Reproductive function in males | Through study completion, an average of 1 year
  Participants: Male athletes (n=16).
  Total and free testosterone levels in the rested and fasted state. Clinically low levels or levels within the lowest quartile of reference range is indicative of hypogonadotropic hypogonadism plus results from outcome 5.
Gastrointestinal function | Day one
  Participants: Elite athletes and controls.
  The LEAF-Q variable regarding gastrointestinal function will be used (se Outcome 5).
Injury | Day one
  Participants: Elite athletes and controls.
  The LEAF-Q variable regarding injury will be used (see Outcome 5).
Self- reported symptoms of depression | Day one
  Participants: Elite athletes and controls.
  Symptoms of depression will be assessed using the Major Depression Index comprising of 10 items that are rated on a 6-point Likert scale from 0 (no time) to 5 (all the time). The total score ranges from 0 to 50 where a higher score reflects more symptoms of depression. Recommended cut-off points are 21 for mild depression, 26 for moderate depression, and 31 for severe depression.
Compulsive exercise | Day one
  Participants: Elite athletes and controls.
  Compulsive exercise will be assessed using the Exercise Addiction Inventory that covers six core symptoms of behavioral addictions. Each item is scored on a Likert-scale from 1 (strongly disagree) to 5 (strongly agree) and a total score of >23 indicates high risk of addiction.
The motivation for behavioral changes | Day one
  Participants: Elite athletes and controls.
  The motivation for behavioral cahnges will be assesed by the Motivation to Change Questionnaire comprising 54 items scored on Likert scales where a higher core indicates poorer ability for behavioral changes.
Psychological flexibility | Day one
  Participants: Elite athletes and controls.
  Psychological flexibility will assessed using the Swedish Acceptance and Action Questionnaire that comprises of 6 items that are scored on a Likert scales (0-6). The higher the score the poorer psychological flexibility.
Changes in immune markers from pre to post exercise | Through study completion, an average of 1 year
  Participants: female athletes (n=28) and male athletes (n=16).
  Inflammatory cytokines and immune components will be assessed in the fasted and rested state and post and exercise test.
Microbiota | Through study completion, an average of 1 year
  Participants: female athletes (n=28) and male athletes (n=16).
  Fecal sample, next-generation sequencing of microbial 16S rRNA genes analyzing bacterial diversity, and composition.
Dietary intake | Through study completion, an average of 1 year
  Participants: female athletes (n=28) and male athletes (n=16).
  A 4-day weighed dietary registration using an electronic kitchen scale and an on-line nutrient program.
Maximal aerobic capacity | Through study completion, an average of 1 year
  Participants: female athletes (n=28) and male athletes (n=16).
  Maximal aerobic capacity (VO2peak) will be assessed by a bicycle ergometer exercise test using a heart rate monitor, an air-tight mask covering the mouth and nose and the Vyntus CPX system.
Explosive lower body power | Through through study completion, an average of 1 year
  Participants: female athletes (n=28) and male athletes (n=16).
  Explosive lower body power will be assessed by a counter movement jumping test.
Whole body strength | Through study completion, an average of 1 year
  Participants: female athletes (n=28) and male athletes (n=16).
  Whole body-strength and force production will be assessed by an isometric mid-thigh pull test.
Muscular power | Through study completion, an average of 1 year
  Participants: female athletes (n=28) and male athletes (n=16).
  Wingate-test (cycles at maximal effort for 30 seconds) will be performed to assess muscular power and anaerobic capacity.
Resting Metabolic Rate | Through study completion, an average of 1 year
  Participants: female athletes (n=28) and male athletes (n=16).
  Resting metabolic rate (kcal/day) will be measured using indirect calometry by a ventilated open hood system (Vyntus CPX).
Body composition | Through study completion, an average of 1 year
  Participants: female athletes (n=28) and male athletes (n=16).
  Fat free mass, fat mass and whole-body, femur and lumbar spine bone mineral density, will be assessed by dual-energy x-ray absorptiometry.
Body weight | Through study completion, an average of 1 year
  Participants: female athletes (n=28) and male athletes (n=16).
  Body mass will be assessed using bioimpedance (Inbody 700)
Body height | Through study completion, an average of 1 year
  Participants: female athletes (n=28) and male athletes (n=16).
  Height will be assessed using a stadiometer.
Glucose levels | Through study completion, an average of 1 year
  Participants: female athletes (n=28) and male athletes (n=16).
  Continuous glucose monitoring using the device by Dexcom.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Melin, PhD, Principal Investigator — Linnaeus University
Locations (1):
- Linnaeus University, Kalmar, Småland, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mountjoy M, Ackerman KE, Bailey DM, Burke LM, Constantini N, Hackney AC, Heikura IA, Melin A, Pensgaard AM, Stellingwerff T, Sundgot-Borgen JK, Torstveit MK, Jacobsen AU, Verhagen E, Budgett R, Engebretsen L, Erdener U. 2023 International Olympic Committee's (IOC) consensus statement on Relative Energy Deficiency in Sport (REDs). Br J Sports Med. 2023 Sep;57(17):1073-1097. doi: 10.1136/bjsports-2023-106994. PMID 37752011
- [Background] Melin A, Tornberg AB, Skouby S, Moller SS, Sundgot-Borgen J, Faber J, Sidelmann JJ, Aziz M, Sjodin A. Energy availability and the female athlete triad in elite endurance athletes. Scand J Med Sci Sports. 2015 Oct;25(5):610-22. doi: 10.1111/sms.12261. Epub 2014 May 30. PMID 24888644
- [Background] Mountjoy M, Sundgot-Borgen JK, Burke LM, Ackerman KE, Blauwet C, Constantini N, Lebrun C, Lundy B, Melin AK, Meyer NL, Sherman RT, Tenforde AS, Klungland Torstveit M, Budgett R. IOC consensus statement on relative energy deficiency in sport (RED-S): 2018 update. Br J Sports Med. 2018 Jun;52(11):687-697. doi: 10.1136/bjsports-2018-099193. No abstract available. PMID 29773536
- [Background] Heikura IA, Uusitalo ALT, Stellingwerff T, Bergland D, Mero AA, Burke LM. Low Energy Availability Is Difficult to Assess but Outcomes Have Large Impact on Bone Injury Rates in Elite Distance Athletes. Int J Sport Nutr Exerc Metab. 2018 Jul 1;28(4):403-411. doi: 10.1123/ijsnem.2017-0313. Epub 2018 Jun 12. PMID 29252050
- [Background] Lundy SD, Sangwan N, Parekh NV, Selvam MKP, Gupta S, McCaffrey P, Bessoff K, Vala A, Agarwal A, Sabanegh ES, Vij SC, Eng C. Functional and Taxonomic Dysbiosis of the Gut, Urine, and Semen Microbiomes in Male Infertility. Eur Urol. 2021 Jun;79(6):826-836. doi: 10.1016/j.eururo.2021.01.014. Epub 2021 Feb 8. PMID 33573862
- [Background] Hackney AC, Lane AR, Register-Mihalik J, O'leary CB. Endurance Exercise Training and Male Sexual Libido. Med Sci Sports Exerc. 2017 Jul;49(7):1383-1388. doi: 10.1249/MSS.0000000000001235. PMID 28195945
- [Background] Logue DM, Madigan SM, Melin A, Delahunt E, Heinen M, Donnell SM, Corish CA. Low Energy Availability in Athletes 2020: An Updated Narrative Review of Prevalence, Risk, Within-Day Energy Balance, Knowledge, and Impact on Sports Performance. Nutrients. 2020 Mar 20;12(3):835. doi: 10.3390/nu12030835. PMID 32245088
- [Background] Konda R, Orikasa S. [Studies on reflux nephropathy, I. Evaluation of renal function by urinary excretion of beta 2-microglobulin]. Nihon Hinyokika Gakkai Zasshi. 1984 Feb;75(2):245-54. No abstract available. Japanese. PMID 6379250
- [Background] Rankin A, O'Donovan C, Madigan SM, O'Sullivan O, Cotter PD. 'Microbes in sport' -The potential role of the gut microbiota in athlete health and performance. Br J Sports Med. 2017 May;51(9):698-699. doi: 10.1136/bjsports-2016-097227. Epub 2017 Jan 25. No abstract available. PMID 28432108
- [Background] Tornberg AB, Melin A, Koivula FM, Johansson A, Skouby S, Faber J, Sjodin A. Reduced Neuromuscular Performance in Amenorrheic Elite Endurance Athletes. Med Sci Sports Exerc. 2017 Dec;49(12):2478-2485. doi: 10.1249/MSS.0000000000001383. PMID 28723842
- [Background] Griffiths MD, Szabo A, Terry A. The exercise addiction inventory: a quick and easy screening tool for health practitioners. Br J Sports Med. 2005 Jun;39(6):e30. doi: 10.1136/bjsm.2004.017020. PMID 15911594
- [Background] Melin A, Tornberg AB, Skouby S, Faber J, Ritz C, Sjodin A, Sundgot-Borgen J. The LEAF questionnaire: a screening tool for the identification of female athletes at risk for the female athlete triad. Br J Sports Med. 2014 Apr;48(7):540-5. doi: 10.1136/bjsports-2013-093240. Epub 2014 Feb 21. PMID 24563388
- [Background] Peman J, Peset V, Salavert M, Carreras C, Esteban G. [Microcytic anemia and coproparasitologic findings in a 3-year-old boy]. Enferm Infecc Microbiol Clin. 1997 Feb;15(2):111-2. No abstract available. Spanish. PMID 9101736
- [Background] Bech P, Timmerby N, Martiny K, Lunde M, Soendergaard S. Psychometric evaluation of the Major Depression Inventory (MDI) as depression severity scale using the LEAD (Longitudinal Expert Assessment of All Data) as index of validity. BMC Psychiatry. 2015 Aug 5;15:190. doi: 10.1186/s12888-015-0529-3. PMID 26242577
- [Background] Lundgren T, Parling T. Swedish Acceptance and Action Questionnaire (SAAQ): a psychometric evaluation. Cogn Behav Ther. 2017 Jun;46(4):315-326. doi: 10.1080/16506073.2016.1250228. Epub 2016 Dec 9. PMID 27931161
- [Background] Gard G, Rivano M, Grahn B. Development and reliability of the Motivation for Change Questionnaire. Disabil Rehabil. 2005 Sep 2;27(17):967-76. doi: 10.1080/09638280500052682. PMID 16096250
- [Background] Vanheest JL, Rodgers CD, Mahoney CE, De Souza MJ. Ovarian suppression impairs sport performance in junior elite female swimmers. Med Sci Sports Exerc. 2014 Jan;46(1):156-66. doi: 10.1249/MSS.0b013e3182a32b72. PMID 23846160
- [Background] Woods AL, Rice AJ, Garvican-Lewis LA, Wallett AM, Lundy B, Rogers MA, Welvaert M, Halson S, McKune A, Thompson KG. The effects of intensified training on resting metabolic rate (RMR), body composition and performance in trained cyclists. PLoS One. 2018 Feb 14;13(2):e0191644. doi: 10.1371/journal.pone.0191644. eCollection 2018. PMID 29444097
- [Background] Loucks AB, Thuma JR. Luteinizing hormone pulsatility is disrupted at a threshold of energy availability in regularly menstruating women. J Clin Endocrinol Metab. 2003 Jan;88(1):297-311. doi: 10.1210/jc.2002-020369. PMID 12519869
- See also: Eating Disorder Examination, EDITION 16.0D, (Fairburn, 2008) — https://www.corc.uk.net/media/1274/ede_rcpsychinformation.pdf
- See also: The REDs Seden project Web Site — https://lnu.se/en/research/research-projects/project-relative-energy-deficiency-in-sports/